CLINICAL TRIAL: NCT03057028
Title: Pilot Study of the Safety and Efficacy of Anakinra in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20005870
Record Dates: First submitted 2016-05-04; First posted 2017-02-17 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Open label treatment with Anakinra
Oversight: Data Monitoring Committee: No

ARMS (1):
- anakinra (Experimental): Patients will be treated with anakinra, injected SQ daily in a dose of 100mg for 14 days. Before and after this intervention, patients will undergo cardiopulmonary exercise testing (as well as echocardiography, EKG analysis, and serologic analysis). Subjects will be assessed for changes in exercise capacity, as determined by peak oxygen uptake and ventilatory efficiency to CO2 production slope.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra
  Other Names: Kineret

SUMMARY:
Pulmonary arterial hypertension (PAH) can result in right ventricular failure and death. Anakinra has been used in patients with left sided heart failure, and the present study looks to determine if anakinra is safe and effective in patients with PAH. To accomplish this goal, we plan to evaluate for exercise improvement (as assessed by cardiopulmonary exercise testing) in 10 patients with PAH on anakinra.

DETAILED DESCRIPTION:
Patients with pulmonary arterial hypertension will undergo cardiopulmonary exercise testing (CPET) at baseline and at 2 weeks. After the initial CPET, all patients will receive anakinra as a daily injection for 2 weeks. Patients will be instructed in the use of anakinra during their initial visit. Our primary outcome will be the difference in the exercise capacity of patients with PAH, as measured by maximal uptake of oxygen on CPET.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* functional class II or III symptoms of right ventricular failure despite optimal PAH therapy
* mean pulmonary artery pressure >25mmHg on previous right heart catheterization
* pulmonary arterial wedge pressure <15mmHg on previous right heart catheterization
* pulmonary vascular resistance >3 wood units on previous right heart catheterization

Exclusion Criteria:

* PAH due to connective tissue disease
* angina or electrocardiograph changes that limit maximum exertion during cardiopulmonary exercise testing or baseline EKG changes that limit the ability to detect ischemia
* recent (<14 days) use of anti-inflammatory drugs (not including NSAIDs), chronic inflammatory disorder, malignancy, active infection, or any comorbidity limiting survival or ability to complete the study
* sever kidney dysfunction (eGFR <30mL/min)
* thrombocytopenia (<50,000/mm3), or neutropenia (absolute neutrophil count <1500/mm3)
* refusal by a woman of childbearing potential to use a medically acceptable form of birth control
* history of hypersensitivity to anakinra or E. coli products
* latex or rubber allergy
* inability to give informed consent
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Change in exercise capacity, as determined by peak oxygen consumption and ventilatory efficiency on cardiopulmonary exercise testing | 14 days

SECONDARY OUTCOMES:
Effect of anakinra on serum high sensitivity C-reactive protein | 14 days
Effect of anakinra on serum NT-pro-BNP. | 14 days
Effect of anakinra on serum interleukin-6 | 14 days
Change in symptoms of heart failure (as assessed by questionnaire with the Duke Activity Status Index and Minnesota Living With Heart Failure Questionnaire). | 14 days
Correlate between biomarkers (serum high sensitivity C reactive protein, interluekin-6, and NT-pro BNP) and measures of exercise capacity (peak oxygen consumption and ventilatory efficiency on cardiopulmonary exercise testing) | 14 days
Number of patients with treatment related adverse events related to anakinra in patients with pulmonary arterial hypertension | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Grinnan, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided